CLINICAL TRIAL: NCT04086550
Title: Randomized, Two-arm, Multicenter Study to Evaluate the Safety and Efficacy of Dura Sealant Patch in Reducing CSF Leakage Following Elective Cranial Surgery
Brief Title: Evaluate the Safety and Efficacy of Dura Sealant Patch in Reducing CSF Leakage Following Elective Cranial Surgery
Acronym: ENCASE-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyganics BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIP-2
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Investigational arm (Experimental): Application of LIQOSEAL after closure of dura mater
  Interventions: Device: LIQOSEAL
- Control arm (Active Comparator): Application of Adherus or DurSeal after closure of dura mater
  Interventions: Device: DuraSeal, Adherus

INTERVENTIONS:
Device: LIQOSEAL — Adjunctive bioresorbable patch
  Arms: Investigational arm
Device: DuraSeal, Adherus — synthetic absorbable sealants
  Arms: Control arm

SUMMARY:
The objective of the study is to clinically assess the safety and effectiveness of LIQOSEAL® as a means of reducing intra- as well as post-operative CSF leakage in patients undergoing elective cranial intradural surgery with a dural closure procedure to show noninferiority compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

pre-operative

1. Subjects who are able to provide written informed consent prior to participating in the clinical investigation.
2. Subjects who are ≥ 18 years old.
3. Subjects who are able to comply with the follow-up or other study requirements.
4. Subjects wo are planned for elective surgery including a trepanation to reach the subdural infratentorial space (with lower limit of incision defined as the lower edge of C2) in whom a dural incision will be closed.
5. Female subjects of child bearing potential must agree to use a form of contraception from the time of signing the informed consent form through 90 days post-surgery.

intra-operative

1. Subjects with surgical wound classification Class I/Clean.
2. Subjects with minimally 5 mm of dural space surrounding dural opening.

Exclusion Criteria:

pre-operative

1. Female subjects who are pregnant or breastfeeding.
2. Subjects with an assumed impaired coagulation due to medication or otherwise.
3. Subjects suspected of an infection requiring antibiotics.
4. Subjects with any type of dural diseases in planned dural closure area.
5. Subjects requiring re-opening of planned surgical area within 90 days after surgery.
6. Subjects with a known allergy to any of the components (Lactide-Caprolactone co-polyester; Butanediol-BDI co-polyurethane; Polyethylene glycol Succinimidyl Gluterate; Disodium hydrogen phosphate or D&C Green No 6) of LIQOSEAL®.
7. Subjects who previously received a LIQOSEAL®.
8. Subjects who previously participated in this study or any investigational drug or device study within 30 days of screening.
9. Subjects with a presence of hydrocephalus.
10. Subjects with contra-indication to MRI [cardiac pacemaker or defibrillator, severe claustrophobia, injured by a metallic object that was not removed, cochlear (ear) implants, metallic implants [e.g. knee replacement].

intra-operative

1. Subjects in whom elevation of PEEP has a potential detrimental effect.
2. Subjects who will require a CSF drain, electrodes or other devices passing the dural layer or extra to intracranial bypass surgery.
3. Subjects who have primary closure of the dura mater with synthetic, nonautologous or autologous material other than galea.
4. Subjects in whom no intra-operative CSF leakage is present after primary closure of the dura mater with elevation of PEEP.
5. Subjects who after primary closure (including galea, if applicable) of the dura mater have a gap > 3 mm.
6. Subjects whom dural opening size including 5 mm margin exceeds patch size (8 x 8 cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Composite endpoint defined as successful dural repair without any of the following compared to the control group: intra-operative CSF leakage percutaneous CSF leak significant pseudomeningocele wound infection | 30 days

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - Stanford University, Palo Alto, California
  - Baptist Health, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Lenox Hill Hospital, New York, New York
  - University of Cincinnatti, Cincinnati, Ohio
  - OHSU, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
- University Hospitals of Innsbruck, Innsbruck, Austria
- University Hospital Gent, Ghent, Belgium
- Germany (2):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - UMM, Mannheim
- Molinette Hospital, Torino, Italy
- Netherlands (2):
  - Elisabeth TweeSteden Ziekenhuis, Tilburg
  - UMCU, Utrecht
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Carlson AP, Slot EMH, van Doormaal TPC; ENCASE II study group; Voormolen EHJ, Dankbaar JW, Depauw P, Brouwers B, Germans MR, Baert E, Vandersteene J, Freyschlag CF, Freyschlag J, Thome C, Zenga F, Penner F, Abdulazim A, Sabel M, Rapp M, Beez T, Zuccarello M, Sauvageau E, Abdullah K, Welch B, Langer D, Ellis J, Dehdashti A, VanGompel J, Bendok B, Chaichana K, Liu J, Dogan A, Lim MK, Hayden MG. Evaluate the safety and efficacy of dura sealant patch in reducing cerebrospinal fluid leakage following elective cranial surgery (ENCASE II): study protocol for a randomized, two-arm, multicenter trial. Trials. 2022 Jul 20;23(1):581. doi: 10.1186/s13063-022-06490-8. PMID 35858894